CLINICAL TRIAL: NCT03510858
Title: Colorectal Cancer Testing in Swiss Primary Care: A Pilot Pragmatic Cluster Randomized Controlled Trial in Quality Circles of Physicians
Brief Title: Randomized Controlled Trial on Colorectal Cancer Screening Among Quality Circles of Primary Care Physicians
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: RCTQC2018
Record Dates: First submitted 2018-04-15; First posted 2018-04-27 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Control Groups; Crossing Over, Genetic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: Multilevel training intervention (intervention group)
- Control group with crossover (Other): Participants in the control group will receive the intervention after 12 months, cross-over design
  Interventions: Other: Multilevel training intervention (control group with crossover)

INTERVENTIONS:
Other: Multilevel training intervention (intervention group) — QC meetings with PCPs in the intervention group to reflect on their CRC screening practices and implement changes in sequential Plan-Do-Check-Act (PDCA) quality improvement cycles. In the first meeting, they will be given evidence summaries on CRC screening, a decision support leaflet designed to help them discuss CRC screening with their patients and a patient decision aid in form of a brochure (Plan-Do). PCPs will receive sample FIT kits recommended for organized screening programs and will be encouraged to offer FIT tests if they have not done so before. In the second QC meeting, PCPs will be shown how to fill out the patient data collection form (Check). The third QC meeting will take place after data collection and analysis. Researchers will present their results to the QCs and PCPs will discuss subsequent steps to improve care (Act). The QC will then repeat one PDCA cycle. The control group will receive the same intervention one year later.
  Arms: Intervention group
Other: Multilevel training intervention (control group with crossover) — The control group will undergo a crossover and receive the same intervention one year after the intervention group. QC meetings with PCPs in the intervention group to reflect on their CRC screening practices and implement changes in sequential Plan-Do-Check-Act (PDCA) quality improvement cycles. In the first meeting, they will be given evidence summaries on CRC screening, a decision support leaflet designed to help them discuss CRC screening with their patients and a patient decision aid in form of a brochure (Plan-Do). PCPs will receive sample FIT kits recommended for organized screening programs and will be encouraged to offer FIT tests if they have not done so before. In the second QC meeting, PCPs will be shown how to fill out the patient data collection form (Check). The third QC meeting will take place after data collection and analysis. Researchers will present their results to the QCs and PCPs will discuss subsequent steps to improve care (Act).
  Arms: Control group with crossover

SUMMARY:
In Switzerland, colorectal cancer (CRC) is the third most common cause of death from cancer with 1600 persons dying from CRC each year. CRC screening can prevent most of these deaths. If screening begins at age 50, with either colonoscopy or faecal immunological test (FIT), the absolute risk of dying from CRC at age 80 can be cut in half. The choice between CRC screening methods can be seen as preference-sensitive condition. FIT can detect CRC at a similar rate as colonoscopy, but cannot detect as many polyps and advanced polyps as colonoscopies. Colonoscopy would seem the best choice for patients who want to reduce their risk of developing CRC or dying from CRC, but colonoscopy is an invasive procedure with rare but serious adverse effects. Patients who choose FIT do not need to prepare their bowels, or take a day off, but instead sample their own stool at home and mail the test to the laboratory. Offering the choice of test might also increase overall screening rates. Guidelines from the US Services Task Force (USPSTF) suggest shared decision making as a method for increasing adherence to screening and elicit patients' preferences for screening options.

Family physicians are recognized as the most trusted professional to discuss CRC screening in Switzerland. However, many primary care physicians (PCPs) appear to prefer colonoscopy over FIT, and the preferred method seems to vary widely between regions. Physician preferences and local medical culture likely determine these choices more than patient preference. It may be possible to reduce the number of PCPs who prescribe only one screening method by encouraging them to diagnose their patient's preferences for screening method. In Switzerland, training PCPs with educational support and decision aids increased the number who intend to prescribe both screening modalities in equal proportions (prescription of both colonoscopy and FIT in equal proportions).

To implement the intervention and determine how and if it changes PCP practice over time, the study will be conducted in quality circles (QCs) of PCPs. QCs are usually groups of 6 to 12 PCPs who meet regularly to reflect on their practice. QCs are a multifaceted, step-based intervention for quality improvement that has gained international traction because they can foster long-lasting behaviour change. In Switzerland, 80% of all PCPs attend QC regularly. Through QCs following the principles of Plan-Do-Check-Act (PDCA) quality improvement cycles, PCPs can find ways to lower structural barriers to screening, assess their screening practices, and give each other feedback.

The study hypothesizes that providing PCPs with evidence summaries on CRC screening, decision aids for patients, and sample FIT tests will increase the number of patients screened for CRC, better balance the selection of screening methods (colonoscopy vs. FIT), increase the proportion of patients with whom PCPs discuss CRC testing, and increase the number of patients who make decision for or against CRC screening.

The outcomes in PCPs of QCs allocated to the intervention group will be compared to those in the control group. The outcomes will be measured through anonymous structured patient data collected on 40 consecutive patients by PCPs and questionnaires filled by PCPs.

To ensure that relevant outcomes important for future implementation and dissemination works are collected, the Reach, Effectiveness, Adoption, Implementation and Maintenance (RE-AIM) framework will be followed for structuring the data collection. The RE-AIM framework helps structure the collection of data on the characteristics of the participants invited who finally participate in the study (Reach), on the integration of the planned intervention in their work (Adoption), on the consistency of implementation of the planned intervention by study participants (Implementation), on the maintenance of the intervention effects over time (Maintenance), and finally, on the effectiveness of the intervention on the planned outcomes (Effectiveness). The RE-AIM criteria are useful for identifying the translatability and public health impact of this intervention, and for making clear to future stakeholders the internal and external validity of study results.

This study will test the benefits of a multilevel training program in participatory medicine designed to help PCPs in Switzerland to better diagnose patient preferences for screening and method of screening method (colonoscopy or FIT) through. If the program is successful it will increase the proportion of patients who can decide to undergo testing or not and with which method. This should increase in number of patients who are screened or intend to be screened for CRC, and thus reduce CRC deaths in the longer term.

ELIGIBILITY:
Inclusion Criteria:

* Physician-level: PCPs of different regions in Switzerland participating in Quality Circles comprising 4 to 19 PCPs and willing to participate in the study
* Patient-level: Three Repeated measures over three years on 40 consecutive patients aged 50 to 75 years old seen in PCP offices over a 2 weeks to 2 months period. Patients will be included if there is a face-to-face consultation billed for at least 5 minutes at the practice.

Exclusion Criteria:

* None except criteria which do not respect inclusion criteria.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients which have been tested for CRC | At 16 months after study begin
  PCPs will systematically collect data from 40 consecutive patients, aged 50 to 75 years

SECONDARY OUTCOMES:
Rate at which PCPs discuss CRC screening with eligible patients (patients not tested in recommended intervals, with no contra-indication for screening) | At 16 months after study begin
  PCPs will systematically collect data from 40 consecutive patients, aged 50 to 75 years
Proportion of patients who were previously tested, plan to be tested or refuse tests | At 16 months after study begin
  PCPs will systematically collect data from 40 consecutive patients, aged 50 to 75 years
Compare proportion of patients who were screened or plan to be screened with colonoscopy vs. FIT | At 16 months after study begin
  PCPs will systematically collect data from 40 consecutive patients, aged 50 to 75 years
Intentions to prescribe tests to screen for CRC | At 16 months after study begin
  A questionnaire filled by each participating PCP
Intention to prescribe colonoscopy vs. FIT within the next 6 months | At 16 months after study begin
  Through a questionnaire filled by each participating PCP

CONTACTS AND LOCATIONS:
Overall Officials: Reto Auer, MD, MAS, Principal Investigator — Institute of Primary Health Care of Bern (BIHAM), University of Bern
Locations (1):
- Institute of Primary Health Care (BIHAM), University of Bern, Bern, Switzerland

REFERENCES:
- [Background] Meester RG, Doubeni CA, Lansdorp-Vogelaar I, Goede SL, Levin TR, Quinn VP, Ballegooijen Mv, Corley DA, Zauber AG. Colorectal cancer deaths attributable to nonuse of screening in the United States. Ann Epidemiol. 2015 Mar;25(3):208-213.e1. doi: 10.1016/j.annepidem.2014.11.011. Epub 2014 Dec 5. PMID 25721748
- [Background] Gigerenzer G. Towards a paradigm shift in cancer screening: informed citizens instead of greater participation. BMJ. 2015 May 5;350:h2175. doi: 10.1136/bmj.h2175. No abstract available. PMID 25943239
- [Background] Schroy PC 3rd, Emmons KM, Peters E, Glick JT, Robinson PA, Lydotes MA, Mylvaganam SR, Coe AM, Chen CA, Chaisson CE, Pignone MP, Prout MN, Davidson PK, Heeren TC. Aid-assisted decision making and colorectal cancer screening: a randomized controlled trial. Am J Prev Med. 2012 Dec;43(6):573-83. doi: 10.1016/j.amepre.2012.08.018. PMID 23159252
- [Background] Salas D, Vanaclocha M, Ibanez J, Molina-Barcelo A, Hernandez V, Cubiella J, Zubizarreta R, Andreu M, Hernandez C, Perez-Riquelme F, Cruzado J, Carballo F, Bujanda L, Sarasqueta C, Portillo I, de la Vega-Prieto M, Morillas JD, Valentin V, Lanas A, Quintero E, Castells A. Participation and detection rates by age and sex for colonoscopy versus fecal immunochemical testing in colorectal cancer screening. Cancer Causes Control. 2014 Aug;25(8):985-97. doi: 10.1007/s10552-014-0398-y. Epub 2014 May 24. PMID 24859111
- [Background] Inadomi JM, Vijan S, Janz NK, Fagerlin A, Thomas JP, Lin YV, Munoz R, Lau C, Somsouk M, El-Nachef N, Hayward RA. Adherence to colorectal cancer screening: a randomized clinical trial of competing strategies. Arch Intern Med. 2012 Apr 9;172(7):575-82. doi: 10.1001/archinternmed.2012.332. PMID 22493463
- [Background] US Preventive Services Task Force; Bibbins-Domingo K, Grossman DC, Curry SJ, Davidson KW, Epling JW Jr, Garcia FAR, Gillman MW, Harper DM, Kemper AR, Krist AH, Kurth AE, Landefeld CS, Mangione CM, Owens DK, Phillips WR, Phipps MG, Pignone MP, Siu AL. Screening for Colorectal Cancer: US Preventive Services Task Force Recommendation Statement. JAMA. 2016 Jun 21;315(23):2564-2575. doi: 10.1001/jama.2016.5989. PMID 27304597
- [Background] Bulliard JL, Ducros C, Levi F. [Organized screening for colorectal cancer: challenges and issues for a Swiss pilot study]. Rev Med Suisse. 2012 Jul 11;8(348):1464-7. French. PMID 22934475
- [Background] Klabunde CN, Lanier D, Nadel MR, McLeod C, Yuan G, Vernon SW. Colorectal cancer screening by primary care physicians: recommendations and practices, 2006-2007. Am J Prev Med. 2009 Jul;37(1):8-16. doi: 10.1016/j.amepre.2009.03.008. Epub 2009 May 13. PMID 19442479
- [Background] McQueen A, Bartholomew LK, Greisinger AJ, Medina GG, Hawley ST, Haidet P, Bettencourt JL, Shokar NK, Ling BS, Vernon SW. Behind closed doors: physician-patient discussions about colorectal cancer screening. J Gen Intern Med. 2009 Nov;24(11):1228-35. doi: 10.1007/s11606-009-1108-4. Epub 2009 Sep 18. PMID 19763699
- [Background] Meissner HI, Breen N, Klabunde CN, Vernon SW. Patterns of colorectal cancer screening uptake among men and women in the United States. Cancer Epidemiol Biomarkers Prev. 2006 Feb;15(2):389-94. doi: 10.1158/1055-9965.EPI-05-0678. PMID 16492934
- [Background] Cooper GS, Koroukian SM. Geographic variation among Medicare beneficiaries in the use of colorectal carcinoma screening procedures. Am J Gastroenterol. 2004 Aug;99(8):1544-50. doi: 10.1111/j.1572-0241.2004.30902.x. PMID 15307875
- [Background] Wennberg JE. Unwarranted variations in healthcare delivery: implications for academic medical centres. BMJ. 2002 Oct 26;325(7370):961-4. doi: 10.1136/bmj.325.7370.961. No abstract available. PMID 12399352
- [Background] Mulley AG, Trimble C, Elwyn G. Stop the silent misdiagnosis: patients' preferences matter. BMJ. 2012 Nov 8;345:e6572. doi: 10.1136/bmj.e6572. No abstract available. PMID 23137819
- [Background] Selby K, Cornuz J, Gachoud D, Bulliard JL, Nichita C, Dorta G, Ducros C, Auer R. Training primary care physicians to offer their patients faecal occult blood testing and colonoscopy for colorectal cancer screening on an equal basis: a pilot intervention with before-after and parallel group surveys. BMJ Open. 2016 May 13;6(5):e011086. doi: 10.1136/bmjopen-2016-011086. PMID 27178977
- [Background] Beyer M, Gerlach FM, Flies U, Grol R, Krol Z, Munck A, Olesen F, O'Riordan M, Seuntjens L, Szecsenyi J. The development of quality circles/peer review groups as a method of quality improvement in Europe. Results of a survey in 26 European countries. Fam Pract. 2003 Aug;20(4):443-51. doi: 10.1093/fampra/cmg420. PMID 12876119
- [Background] Rohrbasser A, Mickan S, Harris J. Exploring why quality circles work in primary health care: a realist review protocol. Syst Rev. 2013 Dec 9;2:110. doi: 10.1186/2046-4053-2-110. PMID 24321626
- [Background] Meyer-Nikolic VA, H.M., Qualitätsentwicklung in der ambulanten Medizin CH: Q-Monitoring-Resultate schaffen Übersicht. Schweizerische Ärztezeitung, 2012. 93.
- [Background] Langley, G.J., et al., The Improvement Guide: A Practical Approach to Enhancing Organizational Performance. 2009: Wiley.
- [Background] Glasgow RE. RE-AIMing research for application: ways to improve evidence for family medicine. J Am Board Fam Med. 2006 Jan-Feb;19(1):11-9. doi: 10.3122/jabfm.19.1.11. PMID 16492000